CLINICAL TRIAL: NCT02437851
Title: A Multicenter Observational and Feasibility Study of Excision of Superficially Invasive Squamous Cell Carcinoma (SISCCA) of the Anal Canal and Perianus in HIV-Infected Persons
Brief Title: Surgery in Treating Patients With Early Stage Anal Canal or Perianal Cancer and HIV Infection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); AIDS and Cancer Specimen Resource (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-092; NCI-2014-02056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-092 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-092 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2015-01-14; First posted 2015-05-08 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Anal Squamous Cell Carcinoma; HIV Infection; Stage 0 Anal Canal Cancer; Stage I Anal Canal Cancer
MeSH Terms: conditions — Anus Neoplasms; HIV Infections; Anal Canal Carcinoma

STUDY DESIGN:
Intervention Model Description: Surgical removal of SISCCA with quarterly monitoring for recurrence and treatment of anal high-grade squamous intraepithelial lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (surgery) (Experimental): Participants undergo therapeutic conventional surgery to remove anal or perianal cancer (SISCCA). Any HSIL remaining is treated with the goal for complete eradication in accordance with clinician and participant preference.
  Interventions: Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Therapeutic Conventional Surgery — Undergo surgery to remove anal or perianal cancer (SISCCA)

SUMMARY:
This phase II trial studies surgery in treating patients with anal canal or perianal cancer that is small and has not spread deeply into the tissues and human immunodeficiency virus (HIV) infection. Local surgery may be a safer treatment with fewer side effects than bigger surgery or radiation and chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of participants who develop treatment failure by 3 years is less than 25%, defined as the occurrence of distant or any nodal metastases or recurrence of cancer requiring chemotherapy (CMT), defined as a cancer that no longer meets the definition of superficially invasive squamous cell carcinoma (SISCCA) or a cancer that cannot be excised with a clear margin or preservation of sphincter function, or those who develop SISCCA recurrence but elect to undergo CMT rather than repeat excision in patients originally treated with excision of anal canal and perianal SISCCA.

II. To define the 1-year proportion of participants who develop incident anal squamous cancers at sites other than the location of the index SISCCA in patients treated with excision of anal canal and perianal SISCCA.

SECONDARY OBJECTIVES:

I. To determine morbidities associated with local excision of SISCCA and treatment of concomitant HSIL, including non-healing ulcer, fissure, persistent pain and bleeding, stricture, incontinence, and colostomy at 3 years after enrollment.

EXPLORATORY OBJECTIVES:

I. To determine the human papillomavirus (HPV) type in cancer and compare to that of overlying high-grade squamous intraepithelial lesions (HSIL) and HSIL biopsies collected concurrently that did not progress to cancer.

II. To determine and compare the HPV integration site in the anal cancer as well as in HSIL overlying or contiguous with the cancer and HSIL biopsies collected concurrently that did not progress to cancer.

III. Perform gene expression array analysis comparing expression in anal cancer with HSIL overlying or contiguous with the cancer.

IV. Perform gene expression array analysis comparing expression in HSIL biopsies that progressed to cancer with non-progressing HSIL biopsies at other locations.

V. Characterize genetic changes in anal cancers compared with HSIL overlying or contiguous with the cancer.

VI. Characterize genetic changes in HSIL biopsies that progressed to cancer compared with non-progressing HSIL biopsies at other locations.

VII. Perform gene expression array analysis and characterize genetic changes of SISCCAs that were cured with wide local excision for comparison with SISCCAs that progressed after wide local excision.

OUTLINE:

Patients undergo surgery to remove anal or perianal cancer. Any HSIL remaining is treated with the goal for complete eradication in accordance with clinician and participant preference.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* A single, biopsy-proven SISCCA as defined by the LAST criteria (=< 3mm depth of invasion, horizontal spread of =< 7 mm, and completely excised with at least 1 mm margin clear of cancer irrespective of the amount of HSIL) documented per investigator assessment in combination with the pathology report within 12 months before Segment B enrollment.
* No evidence of any lymph node spread or distant metastases as determined by PET CT imaging within 16 weeks before Segment B enrollment. Alternatively, for those without PET CT capability, an MRI or CT of the abdomen and pelvis and a chest x-ray confirming no evidence of metastatic disease is acceptable.
* Clinician believes that eradication of concomitant HSIL is reasonable and feasible based on the extent of disease and overall medical condition of the subject
* HIV-1 infection, as documented by one of the following: licensed HIV screening (antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay, Documentation of HIV diagnosis in the medical record by a licensed HIV rapid test health care provider, HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL, or Documentation of receipt of ART by a licensed health care provider.
* Prior to Segment B enrollment, patients on combination anti-retroviral therapy (cART) will be required to have a minimum cluster of differentiation (CD)4 count of >= 200 and patients not on cART will be required to have a minimum CD4 count of >=350 to be eligible for the study; patients not currently on cART who have a CD4 count > 200 and who agree to start cART immediately will be eligible for participation; laboratory data should be obtained within 16 weeks prior to Segment B enrollment
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Participants must have a life expectancy of 2 years or more
* Participants must not have any other concurrent malignancy
* Participants must be age 18 years old or older.
* Leukocytes: >= 3,000/mm^3
* Absolute neutrophil count: >= 1,500/mm^3
* Platelets: >= 100,000/mm^3
* Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to randomization enrollment; female participants enrolled in the treatment arm are advised to not become pregnant during study participation; all women of childbearing potential must agree to either commit to continued abstinence from heterosexual intercourse or use a reliable birth control method (oral contraceptive pills, intrauterine device, Nexplanon, DepoProvera, or bilateral tubal ligation, etc., or another acceptable method as determined by the investigator) during the entire period of the trial (5 years or more), and must not intend to become pregnant during study participation and for 3 months after treatment is discontinued if the participant is enrolled in the treatment arm.
* Men should not father a child while in this study; men who could father a child must agree to use at least one form of birth control or continued abstinence from heterosexual intercourse if receiving topical treatment during during the study and for 2 weeks after stopping topical treatment
* Participants must be able to understand and willing to sign a written informed consent document
* Participants must, in the opinion of the Investigator, be capable of complying with the requirements of this protocol

Exclusion Criteria:

* Anal cancer that cannot be completely excised with a >=1 mm clear margin from surrounding tissue or where excision to obtain a clear margin would compromise sphincter function or anal canal diameter
* Concurrent anal canal or perianal HSIL or condyloma that in the judgment of the clinician cannot be cleared or can only be cleared with undue morbidity to the patient
* No prior history of anal cancer, including SISCCA
* Ongoing use of anticoagulant therapy other than aspirin or non-steroidal anti-inflammatory drugs (NSAIDS) that cannot be stopped for surgical procedures
* Acute treatment for an infection (excluding fungal infection of the skin and sexually transmitted infections) or other serious medical illness within 2 weeks before enrollment
* Current systemic chemotherapy or radiation therapy that potentially causes bone marrow suppression that would preclude safe treatment of HSIL; Note: Kaposi's sarcoma limited to the skin is not exclusionary unless requiring systemic chemotherapy
* The participant's SISCCA must not have been ablated.
* Participants who are receiving any other investigational agents within 4 weeks prior to enrollment. Investigational antiretroviral agents for HIV are acceptable.
* Participant plans to relocate away from the study site during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
To determine if the proportion of participants who develop treatment failure by 3 years is less than 25%. | 3 years after surgery to remove SISCCA
  Treatment failure is specifically defined as the occurrence of distant or any nodal metastases or recurrence of cancer that no longer meets the definition of SISCCA and that cannot be excised with a clear margin or preservation of sphincter function and requires CMT, or those who develop SISCCA recurrence but elect to undergo CMT rather than repeat excision in patients originally treated with excision of anal canal and perianal SISCCA.

SECONDARY OUTCOMES:
The cumulative proportion of study participants who have experienced treatment failure by 3 years will be estimated using the product-limit estimate and its 95% confidence interval using Greenwood's formula. | 3 years after surgery to remove SISCCA
  To determine morbidities associated with local excision of SISCCA and treatment of concomitant HSIL
The rate of treatment related adverse events including non-healing ulcer, fissure, persistent pain and bleeding, stricture, incontinence, and colostomy 6 months after excision of SISCCA. | 6 months after surgery to remove SISCCA
  To determine morbidities associated with local excision of SISCCA and treatment of concomitant HSIL

OTHER OUTCOMES:
Collection of clinical specimens (composite) | Up to 36 months
  Clinical specimens, specifically the index SISCCA and the overlying or adjacent HSIL, and HSIL that did not progress to SISCCA and other clinical data will be collected to create a bank of well-annotated specimens that will enable correlative science: to assess viral factors in HSIL progression to cancer and to identify host factors in HSIL progression to cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Goldstone, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Grady Health System, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Laser Surgery Care, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fuchshuber PR, Rodriguez-Bigas M, Weber T, Petrelli NJ. Anal canal and perianal epidermoid cancers. J Am Coll Surg. 1997 Nov;185(5):494-505. doi: 10.1016/s1072-7515(97)00094-x. PMID 9358099
- [Background] Steele SR, Varma MG, Melton GB, Ross HM, Rafferty JF, Buie WD; Standards Practice Task Force of the American Society of Colon and Rectal Surgeons. Practice parameters for anal squamous neoplasms. Dis Colon Rectum. 2012 Jul;55(7):735-49. doi: 10.1097/DCR.0b013e318255815e. No abstract available. PMID 22706125
- [Background] Benson AB, Venook AP, Al-Hawary MM, Cederquist L, Chen YJ, Ciombor KK, Cohen S, Cooper HS, Deming D, Engstrom PF, Garrido-Laguna I, Grem JL, Grothey A, Hochster HS, Hoffe S, Hunt S, Kamel A, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Murphy JD, Nurkin S, Saltz L, Sharma S, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Wuthrick E, Gregory KM, Freedman-Cass DA. NCCN Guidelines Insights: Colon Cancer, Version 2.2018. J Natl Compr Canc Netw. 2018 Apr;16(4):359-369. doi: 10.6004/jnccn.2018.0021. PMID 29632055
- [Background] Leonard D, Beddy D, Dozois EJ. Neoplasms of anal canal and perianal skin. Clin Colon Rectal Surg. 2011 Mar;24(1):54-63. doi: 10.1055/s-0031-1272824. PMID 22379406
- [Background] Oehler-Janne C, Huguet F, Provencher S, Seifert B, Negretti L, Riener MO, Bonet M, Allal AS, Ciernik IF. HIV-specific differences in outcome of squamous cell carcinoma of the anal canal: a multicentric cohort study of HIV-positive patients receiving highly active antiretroviral therapy. J Clin Oncol. 2008 May 20;26(15):2550-7. doi: 10.1200/JCO.2007.15.2348. Epub 2008 Apr 21. PMID 18427149
- [Background] Wexler A, Berson AM, Goldstone SE, Waltzman R, Penzer J, Maisonet OG, McDermott B, Rescigno J. Invasive anal squamous-cell carcinoma in the HIV-positive patient: outcome in the era of highly active antiretroviral therapy. Dis Colon Rectum. 2008 Jan;51(1):73-81. doi: 10.1007/s10350-007-9154-7. Epub 2007 Dec 8. PMID 18066626
- [Background] Darragh TM, Colgan TJ, Cox JT, Heller DS, Henry MR, Luff RD, McCalmont T, Nayar R, Palefsky JM, Stoler MH, Wilkinson EJ, Zaino RJ, Wilbur DC; Members of LAST Project Work Groups. The Lower Anogenital Squamous Terminology Standardization Project for HPV-Associated Lesions: background and consensus recommendations from the College of American Pathologists and the American Society for Colposcopy and Cervical Pathology. J Low Genit Tract Dis. 2012 Jul;16(3):205-42. doi: 10.1097/LGT.0b013e31825c31dd. PMID 22820980
- [Background] Beahrs OH, Wilson SM. Carcinoma of the anus. Ann Surg. 1976 Oct;184(4):422-8. doi: 10.1097/00000658-197610000-00004. PMID 189707
- [Background] Klas JV, Rothenberger DA, Wong WD, Madoff RD. Malignant tumors of the anal canal: the spectrum of disease, treatment, and outcomes. Cancer. 1999 Apr 15;85(8):1686-93. doi: 10.1002/(sici)1097-0142(19990415)85:83.0.co;2-7. PMID 10223561
- [Background] Chang GJ, Berry JM, Jay N, Palefsky JM, Welton ML. Surgical treatment of high-grade anal squamous intraepithelial lesions: a prospective study. Dis Colon Rectum. 2002 Apr;45(4):453-8. doi: 10.1007/s10350-004-6219-8. PMID 12006924
- [Background] Pineda CE, Berry JM, Jay N, Palefsky JM, Welton ML. High-resolution anoscopy targeted surgical destruction of anal high-grade squamous intraepithelial lesions: a ten-year experience. Dis Colon Rectum. 2008 Jun;51(6):829-35; discussion 835-7. doi: 10.1007/s10350-008-9233-4. Epub 2008 Mar 25. PMID 18363070
- [Background] Zilli T, Schick U, Ozsahin M, Gervaz P, Roth AD, Allal AS. Node-negative T1-T2 anal cancer: radiotherapy alone or concomitant chemoradiotherapy? Radiother Oncol. 2012 Jan;102(1):62-7. doi: 10.1016/j.radonc.2011.09.015. Epub 2011 Oct 10. PMID 21993403
- [Background] Ortholan C, Ramaioli A, Peiffert D, Lusinchi A, Romestaing P, Chauveinc L, Touboul E, Peignaux K, Bruna A, de La Roche G, Lagrange JL, Alzieu C, Gerard JP. Anal canal carcinoma: early-stage tumors < or =10 mm (T1 or Tis): therapeutic options and original pattern of local failure after radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):479-85. doi: 10.1016/j.ijrobp.2004.09.060. PMID 15890590
- [Background] Ortholan C, Resbeut M, Hannoun-Levi JM, Teissier E, Gerard JP, Ronchin P, Zaccariotto A, Minsat M, Benezery K, Francois E, Salem N, Ellis S, Azria D, Champetier C, Gross E, Cowen D. Anal canal cancer: management of inguinal nodes and benefit of prophylactic inguinal irradiation (CORS-03 Study). Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1988-95. doi: 10.1016/j.ijrobp.2011.02.010. Epub 2011 May 11. PMID 21570207
- [Background] Goldstone SE, Hundert JS, Huyett JW. Infrared coagulator ablation of high-grade anal squamous intraepithelial lesions in HIV-negative males who have sex with males. Dis Colon Rectum. 2007 May;50(5):565-75. doi: 10.1007/s10350-006-0874-x. PMID 17380365
- [Background] Goldstone RN, Goldstone AB, Russ J, Goldstone SE. Long-term follow-up of infrared coagulator ablation of anal high-grade dysplasia in men who have sex with men. Dis Colon Rectum. 2011 Oct;54(10):1284-92. doi: 10.1097/DCR.0b013e318227833e. PMID 21904144
- [Background] Stier EA, Goldstone SE, Berry JM, Panther LA, Jay N, Krown SE, Lee J, Palefsky JM. Infrared coagulator treatment of high-grade anal dysplasia in HIV-infected individuals: an AIDS malignancy consortium pilot study. J Acquir Immune Defic Syndr. 2008 Jan 1;47(1):56-61. doi: 10.1097/QAI.0b013e3181582d93. PMID 18156992
- [Background] Marks DK, Goldstone SE. Electrocautery ablation of high-grade anal squamous intraepithelial lesions in HIV-negative and HIV-positive men who have sex with men. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):259-65. doi: 10.1097/QAI.0b013e3182437469. PMID 22134151
- [Background] Goldstone SE, Johnstone AA, Moshier EL. Long-term outcome of ablation of anal high-grade squamous intraepithelial lesions: recurrence and incidence of cancer. Dis Colon Rectum. 2014 Mar;57(3):316-23. doi: 10.1097/DCR.0000000000000058. PMID 24509453
- [Background] FALKSON G, SCHULZ EJ. Skin changes in patients treated with 5-fluorouracil. Br J Dermatol. 1962 Jun;74:229-36. doi: 10.1111/j.1365-2133.1962.tb13497.x. No abstract available. PMID 13891467
- [Background] Maiman M, Watts DH, Andersen J, Clax P, Merino M, Kendall MA. Vaginal 5-fluorouracil for high-grade cervical dysplasia in human immunodeficiency virus infection: a randomized trial. Obstet Gynecol. 1999 Dec;94(6):954-61. doi: 10.1016/s0029-7844(99)00407-x. PMID 10576182
- [Background] Brodman M, Dottino P, Friedman F Jr, Heller D, Bleiweiss I, Sperling R. Human papillomavirus-associated lesions of the vagina and cervix. Treatment with a laser and topical 5-fluorouracil. J Reprod Med. 1992 May;37(5):453-6. PMID 1324311
- [Background] Richel O, Wieland U, de Vries HJ, Brockmeyer NH, van Noesel C, Potthoff A, Prins JM, Kreuter A. Topical 5-fluorouracil treatment of anal intraepithelial neoplasia in human immunodeficiency virus-positive men. Br J Dermatol. 2010 Dec;163(6):1301-7. doi: 10.1111/j.1365-2133.2010.09982.x. Epub 2010 Nov 4. PMID 20716208
- [Background] Richel O, de Vries HJ, van Noesel CJ, Dijkgraaf MG, Prins JM. Comparison of imiquimod, topical fluorouracil, and electrocautery for the treatment of anal intraepithelial neoplasia in HIV-positive men who have sex with men: an open-label, randomised controlled trial. Lancet Oncol. 2013 Apr;14(4):346-53. doi: 10.1016/S1470-2045(13)70067-6. Epub 2013 Mar 15. PMID 23499546
- [Background] Graham BD, Jetmore AB, Foote JE, Arnold LK. Topical 5-fluorouracil in the management of extensive anal Bowen's disease: a preferred approach. Dis Colon Rectum. 2005 Mar;48(3):444-50. doi: 10.1007/s10350-004-0901-8. PMID 15747068
- [Background] Mathiesen O, Buus SK, Cramers M. Topical imiquimod can reverse vulvar intraepithelial neoplasia: a randomised, double-blinded study. Gynecol Oncol. 2007 Nov;107(2):219-22. doi: 10.1016/j.ygyno.2007.06.003. Epub 2007 Jul 25. PMID 17655918
- [Background] van Seters M, van Beurden M, de Craen AJ. Is the assumed natural history of vulvar intraepithelial neoplasia III based on enough evidence? A systematic review of 3322 published patients. Gynecol Oncol. 2005 May;97(2):645-51. doi: 10.1016/j.ygyno.2005.02.012. PMID 15863172
- [Background] Poluri RM, Higgins SP. Successful treatment of penile Bowen's disease with 5% imiquimod cream. Int J STD AIDS. 2005 Sep;16(9):649. doi: 10.1258/0956462054944444. No abstract available. PMID 16176641
- [Background] Ramoni S, Cusini M, Gaiani F, Arancio L, Alessi E. Penile intraepithelial carcinoma treated with imiquimod 1% in an HIV-positive patient. J Dermatolog Treat. 2009;20(3):177-8. doi: 10.1080/09546630802562435. No abstract available. PMID 19016064
- [Background] Kreuter A, Hochdorfer B, Stucker M, Altmeyer P, Weiland U, Conant MA, Brockmeyer NH. Treatment of anal intraepithelial neoplasia in patients with acquired HIV with imiquimod 5% cream. J Am Acad Dermatol. 2004 Jun;50(6):980-1. doi: 10.1016/j.jaad.2003.12.025. No abstract available. PMID 15153912
- [Background] Wagstaff AJ, Perry CM. Topical imiquimod: a review of its use in the management of anogenital warts, actinic keratoses, basal cell carcinoma and other skin lesions. Drugs. 2007;67(15):2187-210. doi: 10.2165/00003495-200767150-00006. PMID 17927284
- [Background] Mahto M, Nathan M, O'Mahony C. More than a decade on: review of the use of imiquimod in lower anogenital intraepithelial neoplasia. Int J STD AIDS. 2010 Jan;21(1):8-16. doi: 10.1258/ijsa.2009.009309. PMID 20029061
- [Background] Kreuter A, Potthoff A, Brockmeyer NH, Gambichler T, Stucker M, Altmeyer P, Swoboda J, Pfister H, Wieland U; German Competence Network HIV/AIDS. Imiquimod leads to a decrease of human papillomavirus DNA and to a sustained clearance of anal intraepithelial neoplasia in HIV-infected men. J Invest Dermatol. 2008 Aug;128(8):2078-83. doi: 10.1038/jid.2008.24. Epub 2008 Feb 14. PMID 18273049
- [Background] Fox PA, Nathan M, Francis N, Singh N, Weir J, Dixon G, Barton SE, Bower M. A double-blind, randomized controlled trial of the use of imiquimod cream for the treatment of anal canal high-grade anal intraepithelial neoplasia in HIV-positive MSM on HAART, with long-term follow-up data including the use of open-label imiquimod. AIDS. 2010 Sep 24;24(15):2331-5. doi: 10.1097/QAD.0b013e32833d466c. PMID 20729710
- [Background] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Background] Schlecht NF, Burk RD, Palefsky JM, Minkoff H, Xue X, Massad LS, Bacon M, Levine AM, Anastos K, Gange SJ, Watts DH, Costa MMD, Chen Z, Bang JY, Fazzari M, Hall C, Strickler HD. Variants of human papillomaviruses 16 and 18 and their natural history in human immunodeficiency virus-positive women. J Gen Virol. 2005 Oct;86(Pt 10):2709-2720. doi: 10.1099/vir.0.81060-0. PMID 16186224
- [Background] Da Costa MM, Hogeboom CJ, Holly EA, Palefsky JM. Increased risk of high-grade anal neoplasia associated with a human papillomavirus type 16 E6 sequence variant. J Infect Dis. 2002 May 1;185(9):1229-37. doi: 10.1086/340125. Epub 2002 Apr 16. PMID 12001039
- [Background] Xi LF, Critchlow CW, Wheeler CM, Koutsky LA, Galloway DA, Kuypers J, Hughes JP, Hawes SE, Surawicz C, Goldbaum G, Holmes KK, Kiviat NB. Risk of anal carcinoma in situ in relation to human papillomavirus type 16 variants. Cancer Res. 1998 Sep 1;58(17):3839-44. PMID 9731493
- [Background] Schmitz M, Driesch C, Jansen L, Runnebaum IB, Durst M. Non-random integration of the HPV genome in cervical cancer. PLoS One. 2012;7(6):e39632. doi: 10.1371/journal.pone.0039632. Epub 2012 Jun 27. PMID 22761851
- [Background] Meyerson M, Gabriel S, Getz G. Advances in understanding cancer genomes through second-generation sequencing. Nat Rev Genet. 2010 Oct;11(10):685-96. doi: 10.1038/nrg2841. PMID 20847746
- [Background] Mine KL, Shulzhenko N, Yambartsev A, Rochman M, Sanson GF, Lando M, Varma S, Skinner J, Volfovsky N, Deng T, Brenna SM, Carvalho CR, Ribalta JC, Bustin M, Matzinger P, Silva ID, Lyng H, Gerbase-DeLima M, Morgun A. Gene network reconstruction reveals cell cycle and antiviral genes as major drivers of cervical cancer. Nat Commun. 2013;4:1806. doi: 10.1038/ncomms2693. PMID 23651994
- [Background] Schwarz JK, Payton JE, Rashmi R, Xiang T, Jia Y, Huettner P, Rogers BE, Yang Q, Watson M, Rader JS, Grigsby PW. Pathway-specific analysis of gene expression data identifies the PI3K/Akt pathway as a novel therapeutic target in cervical cancer. Clin Cancer Res. 2012 Mar 1;18(5):1464-71. doi: 10.1158/1078-0432.CCR-11-2485. Epub 2012 Jan 10. PMID 22235101
- [Background] Wingo SN, Gallardo TD, Akbay EA, Liang MC, Contreras CM, Boren T, Shimamura T, Miller DS, Sharpless NE, Bardeesy N, Kwiatkowski DJ, Schorge JO, Wong KK, Castrillon DH. Somatic LKB1 mutations promote cervical cancer progression. PLoS One. 2009;4(4):e5137. doi: 10.1371/journal.pone.0005137. Epub 2009 Apr 2. PMID 19340305
- [Background] Heselmeyer K, du Manoir S, Blegen H, Friberg B, Svensson C, Schrock E, Veldman T, Shah K, Auer G, Ried T. A recurrent pattern of chromosomal aberrations and immunophenotypic appearance defines anal squamous cell carcinomas. Br J Cancer. 1997;76(10):1271-8. doi: 10.1038/bjc.1997.547. PMID 9374370
- [Background] Heselmeyer K, Macville M, Schrock E, Blegen H, Hellstrom AC, Shah K, Auer G, Ried T. Advanced-stage cervical carcinomas are defined by a recurrent pattern of chromosomal aberrations revealing high genetic instability and a consistent gain of chromosome arm 3q. Genes Chromosomes Cancer. 1997 Aug;19(4):233-40. PMID 9258658
- [Background] Heselmeyer K, Schrock E, du Manoir S, Blegen H, Shah K, Steinbeck R, Auer G, Ried T. Gain of chromosome 3q defines the transition from severe dysplasia to invasive carcinoma of the uterine cervix. Proc Natl Acad Sci U S A. 1996 Jan 9;93(1):479-84. doi: 10.1073/pnas.93.1.479. PMID 8552665
- [Background] Gagne SE, Jensen R, Polvi A, Da Costa M, Ginzinger D, Efird JT, Holly EA, Darragh T, Palefsky JM. High-resolution analysis of genomic alterations and human papillomavirus integration in anal intraepithelial neoplasia. J Acquir Immune Defic Syndr. 2005 Oct 1;40(2):182-9. doi: 10.1097/01.qai.0000179460.61987.33. PMID 16186736
- [Background] Deshmukh AA, Suk R, Shiels MS, Sonawane K, Nyitray AG, Liu Y, Gaisa MM, Palefsky JM, Sigel K. Recent Trends in Squamous Cell Carcinoma of the Anus Incidence and Mortality in the United States, 2001-2015. J Natl Cancer Inst. 2020 Aug 1;112(8):829-838. doi: 10.1093/jnci/djz219. PMID 31742639
- [Background] Shiels MS, Pfeiffer RM, Chaturvedi AK, Kreimer AR, Engels EA. Impact of the HIV epidemic on the incidence rates of anal cancer in the United States. J Natl Cancer Inst. 2012 Oct 17;104(20):1591-8. doi: 10.1093/jnci/djs371. Epub 2012 Oct 5. PMID 23042932
- [Background] Chai CY, Tran Cao HS, Awad S, Massarweh NN. Management of Stage I Squamous Cell Carcinoma of the Anal Canal. JAMA Surg. 2018 Mar 1;153(3):209-215. doi: 10.1001/jamasurg.2017.3151. PMID 29049547
- See also: SEER Cancer Stat Facts: Anal Cancer. National Cancer Institute, Bethesda, MD — https://seer.cancer.gov/statfacts/html/anus.html